CLINICAL TRIAL: NCT03049410
Title: A Phase III Multicentre Randomised Controlled Trial to Compare the Efficacy of Robotically Assisted Radical Cystectomy (RARC) and Intracorporeal Urinary Diversion With Open Radical Cystectomy (ORC) in Patients With Bladder Cancer
Brief Title: Trial to Compare Robotically Assisted Radical Cystectomy With Open Radical Cystectomy
Acronym: iROC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/0584
Record Dates: First submitted 2017-02-02; First posted 2017-02-10 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Bladder Cancer
Keywords: Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iRARC (Active Comparator): Intracorporeal Robot Assisted Radical Cystectomy
  Interventions: Procedure: Intracorporeal Robot Assisted Radical Cystectomy
- Open Radical Cystectomy (ORC) (Active Comparator): Open Radical Cystectomy
  Interventions: Procedure: Open Radical Cystectomy

INTERVENTIONS:
Procedure: Intracorporeal Robot Assisted Radical Cystectomy — Intracorporeal robot assisted radical cystoprostatectomy or anterior exenteration
  Arms: iRARC
Procedure: Open Radical Cystectomy — Removal of bladder and adjacent organs
  Arms: Open Radical Cystectomy (ORC)

SUMMARY:
This is a prospective multicentre randomised controlled trial comparing the outcomes from Intracorporeal RARC (iRARC) with open radical cystectomy (ORC) in patients with bladder cancer. The study will recruit patients with non-muscle invasive bladder cancer (NMIBC) or muscle invasive bladder cancer (MIBC) who have selected radical cystectomy for the treatment of bladder cancer. The time of interest for measurement of the primary outcomes will be 90 days post-surgery.

Eligible patients will include those receiving neo-adjuvant chemotherapy (typically gemcitabine and cisplatin) and those having either an ileal conduit or a neo-bladder reconstruction.

Patients who have selected radical cystectomy after appropriate counselling and following a specialist multi-disciplinary team (SMDT) recommendation, will be approached and asked to consent for this study.

Consenting participants will be randomised 1:1 to either iRARC or ORC. Patients will be followed for a minimum of 90 days post-surgery.

The study will be conducted in National Health Service (NHS) Trusts designated as Cancer Centres.

Patients will be stratified by

* Type of urinary diversion (Continent diversion or ileal conduit)
* Performance status
* Centre Trial assessments will be conducted at baseline (before surgery), whilst participants are on admission and then 5, 12, 26 weeks,1 year and 18 months post surgery.

DETAILED DESCRIPTION:
Radical cystectomy (RC) represents the gold standard treatment for invasive bladder cancer. Reductions in morbidity and mortality from this operation have occurred in recent years through refined anaesthesia, surgical techniques, and centralization of services in high volume centres. The multimodal concept of enhanced recovery after RC (ERAS), which includes pre, intra and post operative steps, has also helped to reduce the length of stay and complications after RC further.

For most abdominal surgery, it is recognized that minimally invasive surgery is less morbid than open surgery, and produces improvements in post-operative recovery without altering the curative nature of the procedure. However, to date, there is little or conflicting evidence of any benefit from minimally invasive surgery over open surgery for RC. This may reflect the complex nature of this procedure (involving surgery to both the urinary and gastro-intestinal tracts), limitations of the current evidence or that there is no benefit. To date, three prospective trials have compared RARC with open RC (ORC). However, each has been limited by sample size and design, or their application of RARC with extra-corporeal reconstruction or have yet to report.

The investigators believe that there are no studies (reported or planned) that have compared optimal RARC (e.g. with intra-corporeal reconstruction) with optimal ORC (e.g. high volume centre using ERAS). In addition, the investigators believe none have adequately assessed the rehabilitation from RC. As such, the investigators now propose a prospective RCT to randomize eligible patients to either ORC or RARC. The investigators will focus upon measures of functional recovery and the return to normal activities.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age.
* Male or female
* Histopathological confirmation of bladder cancer (UCC, SCC, adenocarcinoma or rare variant)
* CIS or stage pTa or pT1 or ≥pT2 or mobile bladder mass on bimanual examination under anaesthesia (see Section 22: Definitions for TNM definitions)
* Node status ≤ N1 on imaging criteria or PET -ve outside pelvis
* ECOG grade 0, 1, 2 or 3
* Able to give informed written consent to participate.

Exclusion Criteria:

* Unwilling to undergo cystectomy.
* Previous abdominal surgery rendering them unsuitable for either iRARC or ORC.
* Patients with upper urinary tract disease
* Concomitant disease that would render the patient unsuitable for the trial
* Pregnant or lactating females
* Previous radiotherapy for bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Days at home within 90 days of the surgery | 90 days post surgery
  To compare the number of days alive and out of hospital within 90 days from surgery.

SECONDARY OUTCOMES:
Difficulties due to health conditions measured using WHODAS version 2.0 | 12 months post surgery
  To assess recovery and complications and the return to normal activities.
Quality of Life measured using EQ-5D-5L Health Questionnaire and EORTC QLQ-C30 version 3. | 12 months post surgery
  To assess recovery and complications and the return to normal activities.

CONTACTS AND LOCATIONS:
Overall Officials: John Kelly, Principal Investigator — University College, London; James Catto, Principal Investigator — University College, London
Locations (8):
- United Kingdom (8):
  - North Bristol NHS Trust, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - St James' University Hospital, Leeds
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's Hospital, London
  - Royal Berkshire Hospital, Reading
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dixon S, Hill H, Flight L, Khetrapal P, Ambler G, Williams NR, Brew-Graves C, Kelly JD, Catto JWF; iROC Study Team. Cost-Effectiveness of Robot-Assisted Radical Cystectomy vs Open Radical Cystectomy for Patients With Bladder Cancer. JAMA Netw Open. 2023 Jun 1;6(6):e2317255. doi: 10.1001/jamanetworkopen.2023.17255. PMID 37389878
- [Derived] Catto JWF, Khetrapal P, Ricciardi F, Ambler G, Williams NR, Al-Hammouri T, Khan MS, Thurairaja R, Nair R, Feber A, Dixon S, Nathan S, Briggs T, Sridhar A, Ahmad I, Bhatt J, Charlesworth P, Blick C, Cumberbatch MG, Hussain SA, Kotwal S, Koupparis A, McGrath J, Noon AP, Rowe E, Vasdev N, Hanchanale V, Hagan D, Brew-Graves C, Kelly JD; iROC Study Team. Effect of Robot-Assisted Radical Cystectomy With Intracorporeal Urinary Diversion vs Open Radical Cystectomy on 90-Day Morbidity and Mortality Among Patients With Bladder Cancer: A Randomized Clinical Trial. JAMA. 2022 Jun 7;327(21):2092-2103. doi: 10.1001/jama.2022.7393. PMID 35569079
- [Derived] Albisinni S, Diamand R, Mjaess G, Aoun F, Assenmacher G, Assenmacher C, Verhoest G, Holz S, Naudin M, Ploussard G, Mari A, Minervini A, Tay A, Issa R, Roumiguie M, Bajeot AS, Simone G, Anceschi U, Umari P, Sridhar A, Kelly J, Hendricksen K, Einerhand S, Sandel N, Sanchez-Salas R, Colomer A, Quackels T, Peltier A, Montorsi F, Briganti A, Teoh JYC, Pradere B, Moschini M, Roumeguere T. Defining the Morbidity of Robot-Assisted Radical Cystectomy with Intracorporeal Urinary Diversion: Adoption of the Comprehensive Complication Index. J Endourol. 2022 Jun;36(6):785-792. doi: 10.1089/end.2021.0843. Epub 2022 May 17. PMID 35109696
- [Derived] Catto JWF, Khetrapal P, Ambler G, Sarpong R, Khan MS, Tan M, Feber A, Dixon S, Goodwin L, Williams NR, McGrath J, Rowe E, Koupparis A, Brew-Graves C, Kelly JD. Robot-assisted radical cystectomy with intracorporeal urinary diversion versus open radical cystectomy (iROC): protocol for a randomised controlled trial with internal feasibility study. BMJ Open. 2018 Aug 8;8(8):e020500. doi: 10.1136/bmjopen-2017-020500. PMID 30093510